CLINICAL TRIAL: NCT02376478
Title: On the Impact of Therapeutic Tumor Necrosis Factor-alpha Inhibition on Anogenital Human Papillomavirus Infection
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Kirnbauer, Prof. Dr., Medical University of Vienna
Other Study IDs: EK208/2009
Record Dates: First submitted 2015-02-19; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Psoriasis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Psoriasis; Inflammatory Bowel Diseases | interventions — Infliximab; Adalimumab; Etanercept; fumaric acid; Mesalamine; Sulfasalazine; purine; Mercaptopurine; Methotrexate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Swab samples to detect mucosal HPV DNA using a FDA-approved Assay (Digene Hybrid Capture 2 kit).
  Cervical PAP smears were collected by cytobrush. Whole blood to obtain peripheral blood mononuclear cells and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- TNF-alpha inhibitors: TNF-alpha Inhibitors: patients with psoriasis or inflammatory bowel diseases under TNF-alpha inhibitor monotherapy
  Interventions: Drug: TNF-alpha inhibitors
- Purine/folic acid analogues: Purine/folic acid analogues: patients with psoriasis or inflammatory bowel diseases receiving monotherapy with purine or folic acid analogues, such as azathioprin, 6-mercaptopurine, or methotrexate
  Interventions: Drug: Purine/folic acid analogues
- Combination therapy: Combination therapy: patients with psoriasis or inflammatory bowel diseases receiving combination therapy with TNF-alpha blocker plus purine or folic acid analogues
  Interventions: Drug: TNF-alpha inhibitors; Drug: Purine/folic acid analogues
- Alternative/no medication: Alternative/no medication: patients with psoriasis or inflammatory bowel diseases receiving alternate therapy, such as phototherapy, fumaric acid, mesalazine, or no medication
  Interventions: Drug: Alternative/no medication; Other: Alternative/no medication

INTERVENTIONS:
Drug: TNF-alpha inhibitors — therapy for at least 6 months
  Other Names: Infliximab, adalimumab, etanercept
  Groups: Combination therapy; TNF-alpha inhibitors
Drug: Alternative/no medication — therapy for at least 6 months or no therapy
  Other Names: fumaric acid, mesalazine, sulfasalazine
  Groups: Alternative/no medication
Other: Alternative/no medication — phototherapy for at least 6 months
  Groups: Alternative/no medication
Drug: Purine/folic acid analogues — therapy for at least 6 months
  Other Names: azathioprin, 6-mercaptopurine, methotrexate
  Groups: Combination therapy; Purine/folic acid analogues

SUMMARY:
In this prospective, open, controlled, cross-sectional observational study patients with psoriasis or IBD, who received either anti-TNF-alpha inhibitors or alternates (purine-, folic acid analogues, phototherapy, fumaric ester, mesalazine) for their underlying disease were included.

Anogenital HPV-induced lesions, mucosal HPV DNA and serological status of mucosal low-risk (HPV6) and high-risk HPV (HPV16, HPV18) were determined.

DETAILED DESCRIPTION:
In this prospective, open, controlled, cross-sectional observational study patients with psoriasis or inflammatory bowel diseases (IBD), who received either Tumor necrosis factor-alpha (TNF-Alpha) inhibitors or alternates (purine-, folic acid analogues, phototherapy, fumaric ester, mesalazine) for their underlying disease were included.

Patients were assigned to the following subgroups according to their current therapy for ≥ 6 months: i) TNF-alpha inhibitor monotherapy; ii) monotherapy with purine or folic acid analogues, such as azathioprin, 6-mercaptopurine, or methotrexate iii) combination therapy with TNF-alpha blocker plus purine or folic acid analogues; iv) alternate therapy, such as phototherapy, fumaric acid, mesalazine. The last group additionally included patients that were without any therapy.

Information about duration and severity of illness, current and former disease-related medical treatment, smoking habits and sexual history with emphasis on preexisting human papillomavirus (HPV) infection, including anogenital warts or previous abnormal cervical cytology, and HPV vaccination status were obtained for each patient.

Swab samples were taken at one time point from the penile shaft and glans of men, the vulva and cervix in women, and the perianal region of both genders.

Detection of mucosal human papillomavirus DNA in the samples was performed using the FDA-approved Digene Hybrid Capture 2 kit.

Cervical Papanicolaou (PAP) smears were collected by cytobrush from female patients at the same time.

Blood for determination of serological status was drawn from each patient and peripheral blood mononuclear cells and serum obtained.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 18-80 years of age with a history of psoriasis or inflammatory bowel diseases, namely Crohn's disease and ulcerative colitis, and
* at least 6 month of continuous treatment regimen.

Exclusion Criteria:

* Pregnant or nursing patients and
* patients with inherited immune disorders, human immunodeficiency virus infection, invasive malignancies or psychomotor retardation and
* patients with psoriasis or inflammatory bowel diseases who had received high-dose corticosteroids during the past 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with psoriasis or inflammatory bowel diseases
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Number of anogenital warts, anogenital HPV DNA positivity and mucosal HPV seropositivity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Kirnbauer, MD, Principal Investigator — Medical University of Vienna